CLINICAL TRIAL: NCT05047250
Title: A Phase III, Single-Arm Multicenter Study of Atezolizumab (Anti-PD-L1 Antibody) in High PD-L1 Expression, Chemotherapy-Naïve Patients With Stage IV Non-Squamous or Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Atezolizumab in High PD-L1 Expression, Chemotherapy-Naïve Patients With Stage IV Non-Squamous or Squamous Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML42606
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Participants will receive IV infusion of atezolizumab on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by investigators.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by investigators.
  Other Names: Tecentriq

SUMMARY:
This is a Phase III, single arm, multicenter study designed to evaluate the efficacy and safety of atezolizumab in high PD-L1 expression, chemotherapy-naïve, without a sensitizing EGFR mutation or ALK translocation patients with stage IV non-squamous or squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 or 1.
* Histologically or cytologically confirmed, Stage IV non-squamous or squamous NSCLC.
* No prior treatment for Stage IV non-squamous or squamous NSCLC.
* Patients who have received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy, or chemo-radiotherapy with curative intent for non-metastatic disease must have experienced a treatment free interval of at least 6 months from enrollment since the last chemotherapy, radiotherapy, or chemo-radiotherapy cycle.
* Tumor TC3 or IC3, as determined by SP142 performed by a central laboratory on previously obtained archival tumor tissue or tissue obtained from a biopsy at screening.
* Measurable disease, as defined by RECIST v1.1.
* Adequate hematologic and end-organ function.
* Life expectancy ≥3 months.
* For women of childbearing potential: agreement to remain abstinent or use contraception, and agreement to refrain from donating.

Exclusion Criteria:

* Known sensitizing mutation in the EGFR gene or ALK fusion oncogene.
* Symptomatic, untreated, or actively progressing CNS metastases.
* Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥2 weeks prior to enrollment.
* Current leptomeningeal disease.
* Uncontrolled tumor-related pain.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
* Uncontrolled or symptomatic hypercalcemia.
* Malignancies other than NSCLC within 5 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome.
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within at least 5 months after the last dose of atezolizumab.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Known allergy or hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation.
* Active or history of autoimmune disease or immune deficiency.
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Positive human immunodeficiency virus (HIV) test result at screening.
* Patients with active hepatitis B or active hepatitis C at screening.
* Active tuberculosis.
* Severe infections within 4 weeks prior to randomization, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Significant cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Atezolizumab initiation to death from any cause (up to approximately 28 months)
  Overall survival (OS) is defined as the time from atezolizumab initiation to death from any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Atezolizumab initiation to the first occurrence of disease progression or death from any cause (whichever occurs first), (up to approximately 28 months)
  Progression-free survival (PFS) is defined as the time from atezolizumab initiation to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by investigators according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1).
OS Rate at 1-Year | Atezolizumab initiation to 1-year
  OS rate at 1-year is defined as the probability of participants who have not experienced death from any cause at 1-year after atezolizumab initiation.
OS Rate at 2-Year | Atezolizumab initiation to 2-year
  OS rate at 2-year is defined as the probability of participants who have not experienced death from any cause at 2-year after atezolizumab initiation.
Objective Response Rate (ORR) | Randomization up to approximately 34 months
  Objective response rate (ORR) is defined as the proportion of participants with a complete response (CR) or partial response (PR), as determined by investigators according to RECIST v1.1.
Duration of Response (DOR) | Randomization up to approximately 34 months
  Duration of response (DOR) is defined as the time from the first occurrence of an objective response to disease progression or death from any cause (whichever occurs first), as determined by investigators according to RECIST v1.1.
Percentage of Participants With Adverse Events | Randomization up to approximately 34 months
  Percentage of participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- China (20):
  - Beijing Tiantan Hospital,Capital Medical University, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - Beijing Chest Hospital, Beijing
  - The Third Xiangya Hospital Of Central South University, Changsha
  - Changzhou First People's Hospital, Changzhou
  - Daping Hospital of Third Military Medical University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Sir Run Run Shaw Hospital Zhejiang University, Hangzhou
  - Anhui Province Cancer Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital Of Jinzhou Medical University, Jinzhou
  - Linyishi Cancer Hospital, Linyi
  - Nanjing Chest Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin Cancer Hospital, Tianjin
  - Tumor Center,Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing